CLINICAL TRIAL: NCT06153953
Title: A Comparative Study Between Vacuum Therapy Dressing and Conventional Dressing in Management of Diabetic Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohsen Ahmed Atta, resident- vascular surgery- sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-23-11-01MS
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator)
  Interventions: Device: vacuum device
- group B (Active Comparator)
  Interventions: Other: conventional dressing therapy

INTERVENTIONS:
Device: vacuum device — use of vacuum device in dressing of diabetic wounds
  Arms: group A
Other: conventional dressing therapy — us of conventional dressing with betadine and iruxol in diabetic wounds
  Arms: group B

SUMMARY:
Diabetes is a global epidemic and a leading cause of death by disease. An estimated 366 million people worldwide had diabetes in 2011.(1).The incidence of diabetic foot ulcers (DFUs) and diabetic complications increases as the age increases.(2).Up to 25% of patients with diabetes will suffer from a foot ulcer during their lifetime. Ulceration is a pivotal factor in the causal pathway to infection and amputation.(3,4).Diabetic foot ulcers (DFUs) are the main cause of hospitalization in diabetic patients and they are considered a worldwide health problem. In recent years, the improvement in diabetes therapy and the reinforcement of guidelines have reduced the amputation rate.(5).The etiology of DFU is complex and rarely unifactorial. In general, foot ulcers are the cumulative result of repetitive trauma that wears a hole in the skin. The triad of neuropathy, foot deformity, and minor considers as the major contributing factors of ulcer development.(6).Vacuum therapy or Negative Pressure Wound Therapy is a technology uses a piece of foam in contact with the wound bed, covered by an occlusive dressing and placed under sub atmospheric pressure.(7).In other words NPWT is a non-invasive therapy system that uses controlled negative pressure using a vacuum device to promote wound healing by removing fluid from open wounds through a sealed dressing or a foam dressing connected to a collection container using sub-atmospheric pressure.(8).The system produces granular tissue that has a characteristic rough appearance. The device can decrease the depth and area of large diabetic foot wounds into a shallow, smaller wound.(8,9).NPWT was first proposed by Argenta and Morykwas in 1997. From then it has been approved as an effective modality of dressing in chronic wounds.(1).NPWT is a safe modality of dressing it has shown a few complications. Minor complications encountered in the vacuum-treated patients : erosion of adjacent tissue due to increased local pressure underneath the tubing ,mild reactions of the peri-wound area (i.e. maceration and eczema) , and sudden increase in body temperature.(10)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diabetic non ischemic wounds which match the criteria suitable for the procedure.

Exclusion Criteria:

* • Patients with chronic limb ischemia non-palpable distal pulsation.

  * Lack of good hemostasis in the wound.
  * Patients with malignant ulcers.
  * Hepatic patients and patients receiving radio or chemotherapy.
  * Wounds over untreated osteomyelitis.
  * Wounds with fistulae to organs or body cavities.
  * Presence of necrotic tissue.
  * Exposed arteries/nerves/anastomotic site/organ

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
duration of healing | 6 months
  healing progress

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Background] Blume PA, Walters J, Payne W, Ayala J, Lantis J. Comparison of negative pressure wound therapy using vacuum-assisted closure with advanced moist wound therapy in the treatment of diabetic foot ulcers: a multicenter randomized controlled trial. Diabetes Care. 2008 Apr;31(4):631-6. doi: 10.2337/dc07-2196. Epub 2007 Dec 27. PMID 18162494
- [Background] Apelqvist J, Armstrong DG, Lavery LA, Boulton AJ. Resource utilization and economic costs of care based on a randomized trial of vacuum-assisted closure therapy in the treatment of diabetic foot wounds. Am J Surg. 2008 Jun;195(6):782-8. doi: 10.1016/j.amjsurg.2007.06.023. Epub 2008 Mar 26. PMID 18355797
- [Background] Armstrong DG, Marston WA, Reyzelman AM, Kirsner RS. Comparative effectiveness of mechanically and electrically powered negative pressure wound therapy devices: a multicenter randomized controlled trial. Wound Repair Regen. 2012 May-Jun;20(3):332-41. doi: 10.1111/j.1524-475X.2012.00780.x. PMID 22564228